CLINICAL TRIAL: NCT00935532
Title: Parallel Group Study to Evaluate the Efficacy and Safety of Exenatide Once-Weekly Injection Compared to Once-Daily Insulin in Type 2 Diabetes Mellitus Treated With Oral Antidiabetic(s)
Brief Title: Study to Evaluate the Efficacy and Safety of Exenatide Once-Weekly Injection Compared to Once-Daily Insulin in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-JE-GWBX
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide once weekly; Byetta; glargine; Lantus; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exenatide once weekly (Experimental)
  Interventions: Drug: exenatide once weekly
- insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: exenatide once weekly — subcutaneous injection, 2.0mg, once a week;
  Arms: exenatide once weekly
Drug: insulin glargine — subcutaneous injection, titrated to achieve fasting serum glucose target, once a day
  Other Names: insulin glargine-Lantus
  Arms: insulin glargine

SUMMARY:
The objectives of this clinical trial are to compare the effects of exenatide once weekly and insulin glargine on blood glucose control, body weight, lipids, safety, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* present with type 2 diabetes mellitus
* HbA1c between 7.1% and 11.0% inclusive
* body mass index (BMI) of >18kg/m2 and <35kg/m2, inclusive
* treated with a stable dose regimen of either of biguanide (BG) alone, BG + thiazolidinedione (TZD), BG + sulfonylurea (SU), or BG + TZD + SU for 90 days prior to study start

Exclusion Criteria:

* Have received chronic (>14 consecutive days) systemic adrenocorticosteroid therapy by oral, intravenous, or intramuscular route or intraarticular steroid injection within 4 weeks prior to study start.
* Have been treated with drugs that promote weight loss within 90 days prior to study start.
* Have been treated with drugs that directly affect gastrointestinal motility for > 21 consecutive days within 90 days prior to study start.
* Have had prior exposure to exenatide BID or QW or participated in the clinical trial of exenatide BID or QW (including the case that the study drug was not administered).
* Have been treated for >2 consecutive weeks with any of the following excluded medications within 90 days prior to study start: Insulin, Dipeptidyl peptidase-4 (DPP-4) inhibitors, GLP-1 analogs
* Have received treatment within 30 days prior to study start drug that has not received regulatory approval for any indication.
* Are currently enrolled in any other clinical study or participated in and completed the clinical study within 30 days prior to study start.
* Have donated blood within 30 days prior to study start.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (22):
- Japan (22):
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukuoka
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Toyama

REFERENCES:
- [Derived] Guja C, Frias JP, Suchower L, Hardy E, Marr G, Sjostrom CD, Jabbour SA. Safety and Efficacy of Exenatide Once Weekly in Participants with Type 2 Diabetes and Stage 2/3 Chronic Kidney Disease. Diabetes Ther. 2020 Jul;11(7):1467-1480. doi: 10.1007/s13300-020-00815-z. Epub 2020 Apr 18. PMID 32306296
- [Derived] Inagaki N, Atsumi Y, Oura T, Saito H, Imaoka T. Efficacy and safety profile of exenatide once weekly compared with insulin once daily in Japanese patients with type 2 diabetes treated with oral antidiabetes drug(s): results from a 26-week, randomized, open-label, parallel-group, multicenter, noninferiority study. Clin Ther. 2012 Sep;34(9):1892-908.e1. doi: 10.1016/j.clinthera.2012.07.007. Epub 2012 Aug 9. PMID 22884767

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Subcutaneous injection, 2.0mg, once a week.
Period: Overall Study
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Started | 215 | 212
Completed | 193 | 201
Not Completed | 22 | 11
Not completed — Adverse Event | 11 | 6
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Subject Decision | 2 | 1
Not completed — Sponsor Decision | 0 | 1
Not completed — Loss Glucose Control | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly | Insulin Glargine | Total
Number analyzed (Participants) | 215 | 212 | 427
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 160 | 156 | 316
  >=65 years | 55 | 56 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.44) | 56.4 (11.16) | 56.8 (10.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 64 | 137
  Male | 142 | 148 | 290
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.51 (0.823) | 8.50 (0.791) | 8.50 (0.806)
Weight [Mean (Standard Deviation); unit: kg] | 69.95 (13.246) | 71.03 (13.932) | 70.49 (13.586)
Background Oral Antidiabetic Agent (OAD) [Number; unit: participants]
  Biguanide (BG) | 145 | 142 | 287
  BG+Thiazolidine Derivative (TZD) | 70 | 70 | 140

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Endpoint (Week 26)
Description: Change in HbA1c from baseline to endpoint (Week 26).
Time Frame: Baseline, Week 26
Population: Statistical analysis of this study was performed for the full analysis set (FAS). FAS consisted of randomized patients who received administration of the study drug at least once and had measurement values after administration. Missing data at endpoint was imputed using last observation carried forward (LOCF) approach.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 214 | 212
percentage of total hemoglobin | -1.11 (0.06) | -0.68 (0.06)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; The expected changes in HbA1c from baseline were considered to be the same between the groups, and the common standard deviation assumed to be 1.2%. Assuming a type I error of 0.025 (one-sided), a power of 0.9 and a noninferiority margin of 0.4%, 191 subjects per group would be necessary to confirm the noninferiority by the two-sample t-test. When the proportion of the subjects missing post-baseline data was assumed to be 10%, the target number of subjects were 420 in total (210 subjects/group); Test type: Non-Inferiority or Equivalence — Noninferiority of exenatide QW to insulin glargine with respect to change in HbA1c was to be concluded if the upper limit of the 95% confidence interval (CI) for the treatment difference was less than 0.4%. Change in HbA1c from baseline to endpoint was analyzed using a LOCF ANCOVA model with treatment, baseline HbA1c stratum (<8.5%, >=8.5%), background OAD, and presence/absence of pretreatment with SU as factors and baseline HbA1c as a covariate; p < .001, ANCOVA — No adjustments for multiplicity will be performed; Least Squares Mean Difference = -0.43, 95% CI 2-sided [-0.59 to -0.26], Standard Error of Mean 0.08

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c<=7%
Description: Percentage of subjects achieving HbA1c <=7.0% (for subjects with HbA1c >7% at baseline)
Time Frame: Baseline, Week 26
Population: FAS Population. Only subjects with baseline HbA1c > target were included in calculation. Missing data at endpoint was imputed using LOCF approach.
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 211 | 210
percentage of subjects | 42.2 | 21.0
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Percentage of subjects achieving HbA1c<=7% at endpoint were compared between treatments using a Cochran-Mantel-Haenszel (CMH) test, in which background OAD and presence/absence of pretreatment with SU served as the stratification factors; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c<=6.5%
Description: Percentage of subjects achieving HbA1c <=6.5% (for subjects with HbA1c >6.5% at baseline)
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 214 | 212
percentage of subjects | 20.6 | 4.2
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Percentage of subjects achieving HbA1c<=6.5% at endpoint were compared between treatments using a CMH test, in which background OAD and presence/absence of pretreatment with SU served as the stratification factors; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change in Fasting Serum Glucose (FSG) From Baseline to Endpoint (Week 26)
Description: Change in FSG (centralized measurement) from baseline to endpoint (Week 26)
Time Frame: Baseline, Week 26
Population: FAS Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 212 | 211
mg/dL | -46.09 (2.40) | -40.82 (2.39)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Change in FSG from baseline to endpoint was analyzed using a LOCF ANCOVA model with treatment, background OAD, and presence/absence of pretreatment with SU as factors and baseline FSG as a covariate; Test type: Superiority or Other; p = 0.103, ANCOVA; Least Squares Mean Difference = -5.28, 95% CI 2-sided [-11.62 to 1.07], Standard Error of Mean 3.23

5. Secondary Outcome: Change in Body Weight From Baseline to Endpoint (Week 26)
Description: Change in Body Weight from baseline to endpoint (Week 26)
Time Frame: Baseline, Week 26
Population: FAS Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 214 | 212
kg | -1.67 (0.17) | 0.34 (0.17)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Change in body weight from baseline to endpoint was analyzed using a LOCF ANCOVA model with treatment, background OAD, and presence/absence of pretreatment with SU as factors and baseline body weight as a covariate; Test type: Superiority or Other; p < .001, ANCOVA; Least Squares Mean Difference = -2.01, 95% CI 2-sided [-2.46 to -1.56], Standard Error of Mean 0.23

6. Secondary Outcome: Change in Total Cholesterol From Baseline to Endpoint (Week 26)
Description: Change in Total Cholesterol from baseline to endpoint (Week 26)
Time Frame: Baseline, Week 26
Population: FAS Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 213 | 212
mg/dL | -14.21 (1.67) | -6.32 (1.67)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Change in total cholesterol from baseline to endpoint was analyzed using a LOCF ANCOVA model with treatment, background OAD, and presence/absence of pretreatment with SU as factors and baseline total cholesterol as a covariate; Test type: Superiority or Other; p < .001, ANCOVA; Least Squares Mean Difference = -7.89, 95% CI 2-sided [-12.33 to -3.45], Standard Error of Mean 2.26

7. Secondary Outcome: Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Endpoint (Week 26)
Description: Change in HDL-C from baseline to endpoint (Week 26)
Time Frame: Baseline, Week 26
Population: FAS Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 213 | 212
mg/dL | -0.99 (0.52) | -0.71 (0.51)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Change in HDL-C from baseline to endpoint was analyzed using a LOCF ANCOVA model with treatment, background OAD, and presence/absence of pre-treatment with SU as factors and baseline HDL-C as a covariate; Test type: Superiority or Other; p = 0.689, ANCOVA; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-1.64 to 1.09], Standard Error of Mean 0.69

8. Secondary Outcome: Ratio of Fasting Triglycerides at Endpoint (Week 26) to Baseline
Description: Ratio of Triglycerides (measured in mg/dL) at endpoint (Week 26) to Baseline. Log(Postbaseline Triglycerides) - log(Baseline Triglycerides); change from baseline to endpoint is presented as ratio of endpoint to baseline.
Time Frame: Baseline, Week 26
Population: FAS Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 213 | 212
ratio | 1.00 (1.02) | 1.00 (1.02)
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Insulin Glargine; Triglycerides data were logarithm-transformed and the change at endpoint to baseline, expressed as the ratio, was analyzed using a LOCF ANCOVA model with treatment, background OAD, and presence/absence of pretreatment with SU as factors and baseline triglycerides as a covariate; Test type: Superiority or Other; p = 0.990, ANCOVA; Geometric Least Squares Mean Ratio = 1.00, 95% CI 2-sided [0.94 to 1.06], Standard Error of Mean 1.03

9. Secondary Outcome: Change in Blood Pressure From Baseline to Endpoint (Week 26)
Description: Change in Blood Pressure from baseline to endpoint (Week 26)
Time Frame: Baseline, Week 26
Population: FAS Population. Missing data at endpoint was imputed using LOCF approach.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 214 | 212
mmHg
  Systolic Blood Pressure | -4.5 (14.04) | -2.6 (14.29)
  Diastolic Blood Pressure | -1.1 (9.25) | -2.5 (8.88)

10. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Major Hypoglycemic Events
Description: Major confirmed hypoglycemia was defined as (1) any event accompanying symptoms consistent with hypoglycemia that resulted in loss of consciousness or seizure but resolved promptly in response to administration of glucagon or (2) glucose, or documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) requiring assistance because of severe impairment in consciousness or motor activity whether or not symptoms of hypoglycemia were felt by the patient. Event rate per subject year was calculated for each subject: (number of events observed from a subject/exposure from a subject)*365.25 where exposure = last postbaseline visit date - baseline visit date. Mean and SE were then derived from FAS.
Time Frame: Baseline to Week 26
Population: FAS Population.
Measure: Mean (Standard Error); unit: events per subject-year
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 215 | 212
events per subject-year | 0.00 (0.00) | 0.00 (0.00)

11. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Minor Hypoglycemic Events
Description: Minor confirmed hypoglycemia was defined as any event a patient felt that he or she was experiencing a sign or symptom associated with hypoglycemia that resolved by self-treatment or on its own, and a concurrent self-monitoring fingerstick blood glucose <3.0 mmol/L (54 mg/dL) and not classified as major hypoglycemia. Event rate per subject year was calculated for each subject: (number of events observed from a subject/exposure from a subject)*365.25 where exposure = last postbaseline visit date - baseline visit date. Mean and SE were then derived from FAS.
Time Frame: Baseline to Week 26
Population: FAS Population.
Measure: Mean (Standard Error); unit: events per subject-year
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Number analyzed (Participants) | 215 | 212
events per subject-year | 0.01 (0.01) | 0.16 (0.13)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 6/215 | 5/212
Other Adverse Events (participants affected / at risk) | 145/215 | 65/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=215) | Insulin Glargine (N=212)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=215) | Insulin Glargine (N=212)
Injection site induration (General disorders) | 58 | 3
Nasopharyngitis (Infections and infestations) | 55 | 45
Nausea (Gastrointestinal disorders) | 27 | 6
Constipation (Gastrointestinal disorders) | 24 | 7
Diarrhoea (Gastrointestinal disorders) | 19 | 5
Induration (General disorders) | 18 | 0
Vomiting (Gastrointestinal disorders) | 18 | 5
Injection site pruritus (General disorders) | 14 | 0
Abdominal discomfort (Gastrointestinal disorders) | 11 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days